CLINICAL TRIAL: NCT00381303
Title: GRACE: An Open-label, Multicenter Trial to Compare the Efficacy, Safety, and Tolerability of PREZISTA (Darunavir)/Ritonavir by Gender and Race, When Administered in Combination With an Individually Optimized Background Regimen Over a 48-week Treatment Period.
Brief Title: GRACE: A Study to Compare the Effectiveness, Safety and Tolerability of PREZISTA (Darunavir)/Ritonavir by Gender and Race When Administered With Other Antiretroviral Medications in Human Immunodeficiency Virus (HIV) Positive Women and Men.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec, Inc (Industry)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011869; TMC114HIV3004
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Results first posted 2010-10-19 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: HIV; Infectious
Keywords: HIV; AIDS; Immunodeficiency Virus, Human; Females; Women; PREZISTA; darunavir; TMC114; Protease Inhibitor
MeSH Terms: conditions — Communicable Diseases; Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 001 (Experimental): darunavir 600mg bid for 48 wks,ritonavir 100mg bid for 48 wks
  Interventions: Drug: darunavir; Drug: ritonavir

INTERVENTIONS:
Drug: darunavir — 600mg bid for 48 wks
Drug: ritonavir — 100mg bid for 48 wks

SUMMARY:
The purpose of this study is to evaluate any differences in the effectiveness, safety, and tolerability of PREZISTA (darunavir; DRV) 600 mg, administered with ritonavir (RTV) 100 mg twice a day on virologic response (defined as a viral load (VL) of < 50 copies/mL) over a 48-week treatment period in HIV-positive women and men. Additional antiretroviral (ARV) agents will also be administered and will be chosen by the Investigator based on resistance testing and prior treatment history (referred to as the Optimized Background Regimen (OBR)).

DETAILED DESCRIPTION:
This is a multi-center, open-label (doctors and patients know which drug is being administered), Phase IIIb clinical trial to evaluate differences in effectiveness, safety, and tolerability of darunavir/ritonavir by sex and/or race over a 48-week treatment period. This study will be conducted in HIV positive women and men who have been treated previously with antiretroviral therapy. This study will enroll 70% women and will be conducted in the U.S., Puerto Rico, Mexico and Canada in approximately 420 patients who will receive darunavir 600 mg and ritonavir 100 mg twice daily. The primary objective of this study is to determine the percentage of patients who achieve virologic response, defined as a viral load (VL) of <50 copies/mL at week 48. Secondary study objectives include comparisons of endpoints between women and men as well as race across multiple parameters including but not limited to change in CD4 count from baseline to week 48, time to loss of virologic response (TLOVR), changes in metabolic parameters (blood chemistry), etc.

Within 4 weeks after the Screening Visit (initial visit with investigator to determine eligibility), the Investigator should have received all data required to determine the patient's eligibility and will construct the individual Optimized Background Regimen (OBR) that will be used during the treatment period in combination with darunavir/ritonavir for those patients enrolled in the study. The OBR will consist of additional antiretroviral (ARV) agents that will also be administered during the study chosen by the Investigator and based on resistance testing and prior treatment history. The study Sponsor will provide the following ARV agents, that may be used as options for the OBR: TMC 125 (investigational non-nucleoside reverse transcriptase inhibitor; NNRTI); Truvada (tenofovir/emtricitabine); Viread (tenofovir); Emtriva (emtricitabine); Zidovudine. Other NRTIs (nucleoside reverse transcriptase inhibitors) or NNRTIs may be used at the discretion of the Investigator, but will not be provided by the Sponsor. The Baseline Visit (Day 1) will be followed by a 48-week treatment period during which patients will be evaluated at Weeks 4, 8, 12, 16, 24, 36, 48 and at a final Follow-Up Visit during Week 52. (total of 10 visits from Screening to final visit). At a number of visits throughout the study, blood samples will be obtained to assess defined laboratory values, safety parameters and to determine concentrations of study drugs darunavir, TMC125 (if applicable) and ritonavir). Patients will be assessed for change in CD4 count and HIV-RNA throughout the study. At each visit, vital signs will be assessed and patients will be asked about any untoward medical occurrences and these will be recorded as adverse events (AEs) and/or HIV-related events. Detailed definitions and reporting procedures for AEs will be provided as part of the protocol. Study patients will receive PREZISTA (darunavir) 600 mg boosted with 100 mg of ritonavir orally (by mouth) twice a day in combination with other antiretroviral drugs for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Plasma HIV-RNA >= 1000 copies/mL
* Must be able to comply with protocol requirements

Exclusion Criteria:

* No prior use of PREZISTA (darunavir), TMC125, enfuvirtide, or tipranavir
* No currently active AIDS defining illness, Category C conditions according to the Center for Disease Control [CDC] Classification System for HIV Infection (1993) with the following exceptions, which must be discussed with the Sponsor prior to enrollment: stable cutaneous Kaposi's Sarcoma, Wasting syndrome due to HIV infection
* Not currently using an investigational drug
* Not pregnant or breastfeeding
* No Grade 3 or 4 laboratory abnormality as defined by DAIDS (Division of AIDS, National Institute of Allergy and Infectious Diseases).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec, Inc. Clinical Trial, Study Director — Tibotec, Inc
Locations (46):
- United States (41):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - Sacramento, California
  - Torrance, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - North Palm Beach, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Port Saint Lucie, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Neptune City, New Jersey
  - Newark, New Jersey
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Harlingen, Texas
  - Houston, Texas
  - Longview, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
- Canada (3):
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Puerto Rico (2):
  - Ponce, PR
  - Rio Piedras

REFERENCES:
- [Derived] Tsoukas C, Gilbert L, Lewis T, Hatzakis G, Falcon R, Mrus J. Improvements in Immune Function and Activation with 48-Week Darunavir/Ritonavir-Based Therapy: GRACE Substudy. ISRN AIDS. 2013 Dec 12;2013:358294. doi: 10.1155/2013/358294. eCollection 2013. PMID 24396625
- [Derived] Smith KY, Garcia F, Kumar P, Currier JS, Ryan R, Falcon R, Mrus J, Squires K. Assessing darunavir/ritonavir-based therapy in a racially diverse population: 48-week outcomes from GRACE. J Natl Med Assoc. 2012 Jul-Aug;104(7-8):366-76. doi: 10.1016/s0027-9684(15)30179-6. PMID 23092052
- [Derived] Currier J, Averitt Bridge D, Hagins D, Zorrilla CD, Feinberg J, Ryan R, Falcon R, Tennenberg A, Mrus J, Squires K; GRACE (Gender, Race, And Clinical Experience) Study Group. Sex-based outcomes of darunavir-ritonavir therapy: a single-group trial. Ann Intern Med. 2010 Sep 21;153(6):349-57. doi: 10.7326/0003-4819-153-6-201009210-00002. PMID 20855799

RESULTS

PARTICIPANT FLOW:
Groups:
- Female: darunavir 600 milligram (mg) twice daily dosing (bid) for 48 weeks administered with ritonavir 100 mg bid for 48 weeks.
- Male: darunavir 600 mg twice bid for 48 weeks administered with ritonavir 100 mg bid for 48 weeks.
Period: Overall Study
Arm/Group | Female | Male
Started | 287 | 142
Completed | 193 | 109
Not Completed | 94 | 33
Not completed — Lost to Follow-up | 25 | 9
Not completed — AE/HIV-related event | 22 | 6
Not completed — Non-Adherence | 13 | 6
Not completed — Withdrawal by Subject | 13 | 6
Not completed — Virologic failure | 6 | 4
Not completed — Ineligible to continue the trial | 2 | 1
Not completed — Pregnancy | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Physician's decision to close the site | 3 | 1
Not completed — Subject moved out of state | 2 | 0
Not completed — Subject taking too many different meds | 1 | 0
Not completed — No virologic response by week 12 | 1 | 0
Not completed — Subject was too busy for appointments | 1 | 0
Not completed — Subject did not continue visits | 1 | 0
Not completed — Subject primary physician's decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Female; Male: darunavir (DRV) 600 mg bid for 48 weeks administered with ritonavir 100 mg bid for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Female | Male | Total
Number analyzed (Participants) | 287 | 142 | 429
Age, Continuous [Median (Full Range); unit: years] | 43 [19 to 78] | 45 [21 to 78] | 43 [19 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287 | 0 | 287
  Male | 0 | 142 | 142
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 191 | 73 | 264
  Caucasian/White | 34 | 31 | 65
  Hispanic | 60 | 36 | 96
  Asian | 0 | 2 | 2
  Other | 2 | 0 | 2
Previous Antiretroviral (ARV) Experience: Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) [Number; unit: participants]
  NNRTI: < 1 drug count | 83 | 32 | 115
  NNRTI: >= 1 drug count | 204 | 110 | 314
Previous ARV experience: Protease inhibitor (PI) [Number; unit: participants]
  PI: <2 | 119 | 50 | 169
  PI: >=2 | 168 | 92 | 260
CD4+ cell count [Median (Full Range); unit: cells/L] | 210 [1 to 868] | 175 [2 to 1125] | 200 [1 to 1125]
Plasma log10 copies/mL VL HIV-1 RNA [Mean (Standard Deviation); unit: copies/mL] | 4.65 (0.883) | 4.73 (0.856) | 4.67 (0.874)
Time since HIV-infection diagnosis [Median (Full Range); unit: years] | 10.78 [0.29 to 27.62] | 11.91 [1.21 to 23.76] | 11.3 [0.29 to 27.62]

OUTCOME MEASURES:

1. Primary Outcome: Number of Viral Load (VL) < 50 HIV-1 RNA Copies/mL (Time to Loss of Virologic Response[TLOVR]) Subjects by Sex
Description: TLOVR - responders/non-responders per FDA TLOVR response algorithm. A subject was considered a responder at that time point and that subsequent. A subject was considered a non-responder at a time point in the following situations: discontinued treatment at that time point, a rebound value at that time point and that subsequent or at that time point and that followed by treatment discontinuation, intermittent missing values were considered a response if the immediately preceding and following visits were a response, rebound at earlier time point, or any new, unplanned ARV except in tolerability
Time Frame: Week 48
Population: Intention to Treat (ITT)
Measure: Number; unit: participants
Arm/Group | Female | Male
Number analyzed (Participants) | 287 | 142
participants | 146 | 83
Statistical Analysis 1: Comparison: Female vs Male; Confidence interval of the difference in proportion of response between two sexes estimated by: * Application of delta method to be obtained Standard Error (SE) * Calculation of lower and upper bound using normal approximation to the difference in response rates; Test type: Non-Inferiority or Equivalence — Test for non-inferiority (Delta=15%); p = 0.30, Regression, Logistic — P-Value for difference (Female - Male): Test for non-inferiority (Delta=15%); Estimates from logistic regression analysis include baseline log10 viral load and baseline CD4 cell count as covariates and gender as a factor; Mean Difference (Final Values) = -9.6, 95% CI 2-sided [-19.85 to 0.68], Standard Error of Mean 0.052

2. Secondary Outcome: Number of VL < 50 HIV-1 RNA Copies/mL (TLOVR) Subjects by Race
Description: Intention to Treat population (ITT)
Time Frame: Week 48
Population: ITT
Measure: Number; unit: participants
Arm/Group | Black | Caucasian | Hispanic | Asian | Other
Number analyzed (Participants) | 264 | 65 | 96 | 2 | 2
participants | 128 | 39 | 59 | 2 | 1

3. Secondary Outcome: Number of Etravirine-TMC125 (ETR) Subgroup- VL < 50 HIV-1 RNA Copies/mL (TLOVR) Subjects
Description: The Etravirine-TMC125 (ETR Subgroup population was defined as all ITT subjects who took at least 1 dose of ETR)
Time Frame: Week 48
Population: ETR Subgroup- Intention to Treat population (ITT)
Measure: Number; unit: participants
Arm/Group | Female | Male | Black | Caucasian | Hispanic | Asian | Other
Number analyzed (Participants) | 119 | 88 | 133 | 34 | 36 | 2 | 2
participants | 69 (0.088) | 54 (0.131) | 74 (0.092) | 21 (0.191) | 25 (0.158) | 2 (0.472) | 1 (-1.73)

4. Secondary Outcome: Descriptive Statistics of [TLOVR Non-virologic Failure (VF) Censored] - VL < 50 HIV-1 RNA by Race
Description: TLOVR non-virologic failure (VF) censored. This imputation method differs from the TLOVR algorithm, because subjects that dropped out for reasons other than virologic failure were censored from the time of discontinuation onwards.
Time Frame: Week 48
Population: TLOVR Non-virologic Failure(VF) Censored
Measure: Number; unit: participants
Arm/Group | Black | Caucasian | Hispanic | Asian | Other
Number analyzed (Participants) | 186 | 50 | 74 | 2 | 1
participants | 128 | 39 | 59 | 2 | 1

5. Secondary Outcome: Descriptive Statistics of ETR Subgroup [TLOVR Non-virologic Failure (VF) Censored] - VL < 50 HIV-1 RNA
Description: The Etravirine-TMC125 (ETR Subgroup population was defined as all ITT subjects who took at least 1 dose of ETR)
  TLOVR non-virologic failure(VF) censored. This imputation method differs from the TLOVR algorithm, because subjects that dropped out for reasons other than virologic failure were censored from the time of discontinuation onwards.
Time Frame: Week 48
Population: Etravirine-TMC125 (ETR) Subgroup [TLOVR Non-virologic Failure (VF) Censored]
Measure: Number; unit: participants
Arm/Group | Female | Male | Black | Caucasian | Hispanic | Asian | Other
Number analyzed (Participants) | 87 | 74 | 102 | 26 | 30 | 2 | 1
participants | 69 | 54 | 74 | 21 | 25 | 2 | 1

6. Secondary Outcome: Descriptive Statistics of Change From Baseline in CD4+ Cell Count Using Observed Values
Description: Observed obsevations have no imputation methods applied.
Time Frame: Baseline, Week 48
Population: ITT
Measure: Mean (Standard Error); unit: x10^6 cells/L
Arm/Group | Female | Male | Black | Caucasian | Hispanic | Asian | Other
Number analyzed (Participants) | 188 | 105 | 173 | 47 | 70 | 2 | 1
x10^6 cells/L | 152 (11.2) | 122 (12.3) | 143 (10.8) | 151 (23.8) | 133 (17.0) | 45 (24.5) | 179

7. Secondary Outcome: Descriptive Statistics of ETR Subgroup - Change From Baseline in CD4+ Cell Using Observed Values
Description: The Etravirine-TMC125 (ETR Subgroup population was defined as all ITT subjects who took at least 1 dose of ETR)
Time Frame: Week 48
Population: Etravirine-TMC125 (ETR Subgroup) Intention to Treat population (ITT)
Measure: Mean (Standard Error); unit: x10^6 cells/L
Arm/Group | Female | Male | Black | Caucasian | Hispanic | Asian | Other
Number analyzed (Participants) | 80 | 67 | 93 | 25 | 26 | 2 | 1
x10^6 cells/L | 136 (15.8) | 108 (15.1) | 135 (13.5) | 111 (26.7) | 98 (29.8) | 45 (24.5) | 179

8. Secondary Outcome: Descriptive Statistics of Change From Baseline in CD4+ Cell Count Using the Imputation Method of Last Observation Carried Forward (LOCF)
Description: Last Observation Carried Forward (LOCF) imputation method applied.
Time Frame: Week 48
Population: ITT LOCF
Measure: Mean (Standard Error); unit: x10^6 cells/L
Arm/Group | Female | Male | Black | Caucasian | Hispanic | Asian | Other
Number analyzed (Participants) | 287 | 142 | 264 | 65 | 96 | 2 | 2
x10^6 cells/L | 112 (8.8) | 103 (11.2) | 109 (8.9) | 110 (20.4) | 109 (13.5) | 45 (24.5) | 138 (41.0)

9. Primary Outcome: Number of TLOVR Non-virologic Failure (VF) Censored - VL < 50 HIV-1 RNA Subjects by Sex
Description: as for outcome 4
Time Frame: Week 48
Population: TLOVR non-virologic failure (VF) censored
Measure: Number; unit: participants
Arm/Group | Female | Male
Number analyzed (Participants) | 200 | 113
participants | 146 | 83

10. Secondary Outcome: Descriptive Statistics of ETR Subgroup - Change From Baseline in CD4+ Cell Count Using the Imputation Method of LOCF
Description: The Etravirine-TMC125 (ETR Subgroup population was defined as all ITT subjects who took at least 1 dose of ETR). The Last Observation Carried Forward (LOCF) imputation method was applied.
Time Frame: Week 48
Population: Etravirine-TMC125 (ETR Subgroup) Intention to Treat population (ITT)
Measure: Mean (Standard Error); unit: x10^6 Cells/L
Arm/Group | Female | Male | Black | Caucasian | Hispanic | Asian | Other
Number analyzed (Participants) | 119 | 88 | 133 | 34 | 36 | 2 | 2
x10^6 Cells/L | 107 (12.7) | 98 (14.0) | 113 (12.1) | 84 (21.7) | 90 (22.6) | 45 (24.5) | 138 (41.0)

ADVERSE EVENTS:
Time Frame: 48 Weeks
Arm/Group | Female | Male
Serious Adverse Events (participants affected / at risk) | 47/287 | 33/142
Other Adverse Events (participants affected / at risk) | 73/287 | 33/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Female (N=287) | Male (N=142)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 2 | 2
Cardiac Failures Congestive (Cardiac disorders) | 1 | 0
Cardiac Tamponade (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 2
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Acquired Oesophageal Web (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gatrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal Ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 4
Multi-Organ Failure (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 2 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 1
Abscess (Infections and infestations) | 1 | 1
Abcess Limb (Infections and infestations) | 1 | 1
Bacterial Pyelonephritis (Infections and infestations) | 2 | 2
Bacterial Sepsis (Infections and infestations) | 1 | 1
Bartonellosis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2
Clostridium Difficile Colitis (Infections and infestations) | 1 | 1
Cytomegalovirus Oesophagitis (Infections and infestations) | 0 | 0
Dengue Fever (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteriris Cryptosporidial (Infections and infestations) | 0 | 1
Gonorrhoea (Infections and infestations) | 1 | 0
Herpes Zoster Ophthalmic (Infections and infestations) | 1 | 0
Lung Infection Pseudomonal (Infections and infestations) | 0 | 1
Meningitis Aseptic (Infections and infestations) | 0 | 0
Meningitis Tuberculous (Infections and infestations) | 1 | 0
Meningitis Viral (Infections and infestations) | 1 | 1
Oesophageal Candidiasis (Infections and infestations) | 1 | 0
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 1 | 4
Pneumonia (Infections and infestations) | 10 | 1
Pneumonia Bacterial (Infections and infestations) | 0 | 1
Pneumonia Legionella (Infections and infestations) | 1 | 0
Rectal Abcess (Infections and infestations) | 0 | 1
Septic Arthritis Staphylococcal (Infections and infestations) | 0 | 1
Sinusitus (Infections and infestations) | 0 | 0
Staphylococcal Abcess (Infections and infestations) | 1 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Viral Infection (Infections and infestations) | 1 | 0
Accidental Overdose (Infections and infestations) | 0 | 1
Operative Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alanine Amino Transferase Increased (Investigations) | 0 | 1
Aspartate Amino Transferase Increased (Investigations) | 1 | 1
Blood Amylase Increased (Investigations) | 0 | 1
Blood Lactic Acid Increased (Investigations) | 0 | 1
Transaminases Increased (Investigations) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0
Anal Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Status Epilepticus (Nervous system disorders) | 0 | 1
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 1
Catatonia (Psychiatric disorders) | 1 | 1
Conversion Disorder (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 1
Dependence (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 2
Major Depression (Psychiatric disorders) | 1 | 1
Suicide Attempt (Psychiatric disorders) | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioneurotic Oedema (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Drug Abuser (Social circumstances) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 2
Haemorrhage (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Vascular Insufficiency (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Female (N=287) | Male (N=142)
Lymphadenopathy (Blood and lymphatic system disorders) | 20 | 8
Diarrhoea (Gastrointestinal disorders) | 47 | 31
Nausea (Gastrointestinal disorders) | 70 | 20
Vomiting (Gastrointestinal disorders) | 33 | 9
Oedema Peripheral (General disorders) | 16 | 6
Pyrexia (General disorders) | 14 | 12
Bronchitis (Infections and infestations) | 18 | 7
Oral Candidiasis (Infections and infestations) | 19 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 30 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 16 | 11
Headache (Nervous system disorders) | 26 | 11
Depression (Psychiatric disorders) | 15 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 5
Rash (Skin and subcutaneous tissue disorders) | 23 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If TTCA does not publish within 12 months after study conclusion or after TTCA confirms there will be no multicenter publication, Institution may publish their results from their site individually, provided TTCA has 60 day review for confidentiality and additional 60 day delay for patent application.